CLINICAL TRIAL: NCT03123744
Title: A Histology-Independent Study of the Cyclin Inhibitor Palbociclib in Patients With Advanced Cancer Harboring Aberrations in the Cyclin Pathway
Brief Title: Histology-Independent Study of Palbociclib in Patients With Advanced Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No study funding available.
Sponsor: Razelle Kurzrock, MD (Other)
Responsible Party: Sponsor-Investigator, Razelle Kurzrock, MD, Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IIT 150729
Record Dates: First submitted 2017-03-03; First posted 2017-04-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Cancer, Advanced
Keywords: Palbociclib; Cyclin Pathway; kinase inhibitor
MeSH Terms: conditions — Neoplasms | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, non-randomized Phase II study of palbociclib in adult subjects with recurrent or refractory advanced cancers with aberration(s) in cyclin (CCN/CDK) signaling. Treatment will consist of daily oral administration of palbociclib in 28-day cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib 125 mg (Experimental): Palbociclib is administered orally at a starting dose of 125 mg/day for three weeks followed by one week off. Study measurements will be obtained at baseline and about every 8 weeks thereafter. Subjects will continue study drug until disease progression or unacceptable toxicity.
  Interventions: Drug: Palbociclib 125mg

INTERVENTIONS:
Drug: Palbociclib 125mg — Palbociclib 125 mg is administered orally at a starting dose of 125 mg/day for three weeks followed by one week off. Study evaluations include physical exams, performance status, vital signs, laboratory blood tests, and radiographic or MRI imaging.
  Other Names: Ibrance®

SUMMARY:
The investigational drug being tested in this study is palbociclib. Palbociclib is considered experimental because it is not approved by the FDA for the treatment of all cancers. Palbociclib is currently approved for use in breast cancer. Palbociclib is a drug belonging to a family of drugs called kinase inhibitors. These drugs slow or stop the activity of particular proteins involved in the growth of human cells and in the abnormal growth of cancer cells. Blocking these proteins may decrease or stop tumor growth. The purpose of this study is to assess the safety of the study drug, to see how well it is tolerated, and also to find a safe dose range of the study drug in patients with specific kinds of tumor genetic changes.

DETAILED DESCRIPTION:
This study proposes to give the cyclin dependent kinase (CDK) inhibitor palbociclib to patients with advanced malignancy harboring cyclin pathway aberrations (CCN/CDK alterations). The investigators study will determine whether cyclin signaling aberrations associate with response to this CDK inhibitor. Once completed, this study will identify subpopulations of patients that would best benefit from CDK inhibitor therapy with palbociclib and suggest directions for future study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Pathologically confirmed advanced or metastatic malignancy characterized by one or more of the following:

   * Subject is intolerant to standard therapy
   * Subject refuses standard therapy
   * Malignancy is refractory to standard therapy
   * Malignancy relapsed after standard therapy
   * Malignancy for which there is no standard therapy that improves survival by at least 3 months.
3. Evaluable tumor(s) with documented alteration(s) in CCN/CDK-related gene(s). The CCN/CDK aberration(s) can be identified at any point in the subject's cancer course. CCN/CDK testing must have been performed in a CLIA-certified laboratory. Amplification(s) and/or mutation frequencies will be defined according to the standard of the test used.
4. ECOG Performance Status 0-2
5. Women of childbearing potential must have a negative baseline blood pregnancy test. Women and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study and for at least 30 days after discontinuation of study drug (the half life of palbociclib is about 27 hours in patients with cancer).
6. Subjects must be off other anti-tumor agents for at least 5 half lives of the agent or 4 weeks from the last day of treatment, whichever is shorter. Endocrine therapies (for example for breast or prostate cancer) and anti-Her2 therapies (for example, trastuzumab or lapatinib) are allowed to continue while on this study.
7. Subjects may not be receiving any other experimental agents.
8. Ability to understand and willingness to sign a written consent document.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Subjects who have not recovered from toxicities as a result of prior anticancer therapy, except alopecia and infertility. Recovery is defined as < Grade 2 severity per Common Terminology Criteria for Adverse Events Version 4.0(1) (CTCAE v4.0) or to their clinical baseline.
3. Inability to swallow pills or determination by the investigator that absorption of oral medication would be impaired.
4. Major surgery (not including placement of central lines) within 3 weeks prior to trial enrollment or planned surgery during the course of this study.
5. Any medical condition which, in the opinion of the investigator, would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Response rates in subjects with advanced cancer and aberrations of cyclin pathway gene(s) who are treated with palbociclib | Every 8 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Radiographic or MRI imaging will be assessed approximately every 8 weeks for disease progression.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Every 2-4 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Complete physical exams will be assessed every 2 to 4 weeks during treatment to evaluate the number of patients with a drug toxicity and disease progression.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Every 2-4 weeks from date of enrollment, assessed up to 36 months.
  Laboratory blood tests will be assessed every 2 to 4 weeks during treatment to evaluate the number of patients for drug toxicity and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lippman, MD, Study Director — UCSD
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No